CLINICAL TRIAL: NCT00266604
Title: TOPAMAX� (Topiramate) Initiated as Monotherapy in Epilepsy (TIME): A Multicenter, Outpatient, Open-Label, Study to Evaluate the Dosing, Effectiveness and Safety of TOPAMAX� as Monotherapy in the Treatment of Epilepsy in Clinical Practice
Brief Title: A Study to Evaluate the Dosing, Effectiveness and Safety of Topiramate for the Treatment of Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002869
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Epilepsy; Seizures; Epilepsies, Partial; Epilepsy, Generalized; Seizures, Tonic-Clonic
Keywords: Epilepsy; seizures; new-onset epilepsy; epilepsy relapse; epilepsy monotherapy
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Partial; Epilepsy, Generalized | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The purpose of this study is to identify patient characteristics (such as baseline seizure frequency) that may predict effective doses of topiramate using just that one drug (monotherapy) as initial therapy for epilepsy. Topiramate is an anti-epileptic drug that is approved for the treatment of epilepsy in adults and children 2 years of age and above.

DETAILED DESCRIPTION:
Any number of factors could affect the dosage needs for an anti-epileptic medication, however, various lines of evidence suggest that characteristics of the patient's epilepsy itself could be important determinants. Baseline (i.e., at the start of the study) patient characteristics, particularly seizure frequency, may predict dosage needs when TOPAMAX® (topiramate) is initiated as monotherapy and titrated to an individualized optimal dose. Topiramate is an anti-epileptic drug that is approved for epilepsy either alone (i.e., monotherapy), or in combination with other anti-epileptic medications, in adults and children 2 years of age and above. This is a multicenter, outpatient, open-label, single-arm study to evaluate the dosing, tolerability, effectiveness and safety of topiramate as initial therapy for epilepsy in clinical practice. Patients who have been identified by their physicians as candidates for initial anti-epileptic monotherapy will be enrolled. Patients will begin therapy with topiramate tablets starting at 50 milligrams per day and be titrated to an individualized optimal dose, up to a maximum of 400 milligrams per day, by the end of week 6. Changes to this schedule will be based on a risk-benefit assessment of the patient's clinical condition by the investigator, such as tolerability, or reaching a stable dose sufficient to control their seizures. Treatment with topiramate will last for a total of 24 weeks. The primary outcome of the study is a comparison of the mean stabilized topiramate dose during the last 28 days of treatment for patients reporting 1 to 3 seizures during the 3 months prior to study entry versus patients reporting more than 3 seizures during the 3 months prior to study entry. The study hypothesis is that the average stabilized dose of topiramate will be lower in patients that have had fewer seizures in the 3 months prior to beginning the study. Topiramate tablets starting at 50 milligrams per day and titrated to an individualized optimal dose, up to a maximum of 400 milligrams per day by the end of week 6. Patients will take topiramate tablets by mouth twice a day (morning and evening) for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients having new-onset epilepsy or epilepsy relapse characterized by partial-onset seizures or primary generalized tonic-clonic seizures
* having at least 1 seizure within the 3 months prior to entry
* who are previously untreated for epilepsy, previously treated for epilepsy, or if currently taking epilepsy medication, must have been taking it for less than 6 weeks
* weighing at least 25 kilograms (approximately 55 pounds)
* if female of childbearing potential, must be using an acceptable method of birth control

Exclusion Criteria:

* Patients who have previously taken topiramate for the treatment of epilepsy
* who are currently taking topiramate for any reason
* having active liver disease
* having a clinically significant medical condition or disease
* women who are pregnant or breastfeeding

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2005-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the mean stabilized topiramate dose during the last 28 days of treatment between patients reporting 1 to 3 seizures versus patients reporting more than 3 seizures, during the 3 months prior to study entry

SECONDARY OUTCOMES:
Influence of other patient characteristics on dose; Proportion of subjects remaining seizure-free; Time to stabilized dose; Reduction in seizure frequency

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Topamax Initiated as Monotherapy in Epilepsy (TIME) CSR — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=496&filename=CR002869_CSR.pdf